CLINICAL TRIAL: NCT02626910
Title: Patient Centered Outcomes Research Institute: Mrs. A and Mr. B
Brief Title: Understanding Disparities in Healthcare and Primary Care Provider Quality
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: AD-12-11-4567
Record Dates: First submitted 2015-11-30; First posted 2015-12-10 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-10

CONDITIONS: Physical Disability
Keywords: Disability; Activity of Daily Living; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Second Life: People with disabilities: People with disabilities recruited from the virtual world, Second life.
- Second Life: People without disabilities: People without disabilities recruited from the virtual world, Second life.
- Second Life: Clinicians: Clinicians recruited from the virtual world, Second life.
- Urban group: People with and without disabilities recruited from an Urban setting.

SUMMARY:
The project proposes to fill gaps in the understanding of disparities in healthcare and primary care provider (PCP) quality from the perspectives of adult Medicare beneficiaries with disabilities compared to those without disabilities. Studies document racial/ethnic, economic, and education-related disparities, but little is known about healthcare disparities related to disability.

DETAILED DESCRIPTION:
BACKGROUND: The project proposes to fill gaps in the understanding of disparities in healthcare and primary care provider (PCP) quality from the perspectives of adult Medicare beneficiaries with disabilities compared to those without disabilities. Studies document racial/ethnic, economic, and education-related disparities, but little is known about healthcare disparities related to disability.

OBJECTIVE: The investigators' goal is to engage stakeholders as peers and partners in the development of an evidence-based Patient-Inspired Surveillance Tool for documenting variations in healthcare and PCP quality and any outcome consequences associated with these variations among people with disabilities (PWD) and people without disabilities (PWOD). The tool is intended to provide guidance on programs and policies to ameliorate disparities, improve function, and enhance autonomy in populations of people.

METHODS: The investigators will explore perceptions about the determinants of healthcare and PCP quality in partnership with stakeholders including PWD, PWOD, family of PWD, and healthcare providers in efforts to better understand underlying determinants of healthcare disparities that might be accelerating clinical deterioration. Applying population weighted data and multi-variable methods to patient information included in the Medicare Current Beneficiary Survey (MCBS), the investigators will determine the presence or absence of perceived problems across 5 healthcare and PCP quality "comparators" and (if present) the magnitude of impact on likelihood of patients' functional improvement, functional decline, institutionalization, or death referenced to no status change by 1, 2, and 3 years. A decade of data from the MCBS (on about 40,000 working age and elderly patients) will be applied to ensure adequate statistical power for comparisons. Stakeholders will help interpret the implications of findings and partner with clinician researchers in building the Tool.

PATIENT OUTCOMES: For aim 2, the outcome will be healthcare and PCP quality across 5 "quality comparators" including patients' perceptions about care coordination and quality, access barriers, technical skills of PCP, interpersonal skills of PCP, and the quality of information provided by PCP. Comparisons will be cross sectional contrasting the proportions of people at each stage of disability referenced to PWOD perceiving lower verses higher quality on each comparator. These 5 comparators will become the exposure for aims 3 and 4.

For aims 3 and 4, the outcome will include "no change" (individual remains at the same Activity of Daily Living (ADL)/Instrumental Activity of Daily Living (IADL) stage), "functional improvement" (recovery to a lower ADL/IADL stage), "functional decline" (deterioration to a higher stage of ADL/IADL limitation), "institutionalization" (long-term nursing home), or "death." Comparison will be longitudinal prediction at 1, 2, and 3 years in contrast to no change according to each comparator.

ELIGIBILITY:
Inclusion Criteria:

* Second Life: People with disabilities - only those with disabilities from Second Life.
* Second Life: People without disabilities - only those without disabilities from Second Life.
* Second Life: clinicians - only clinicians from Second Life.
* Urban: either those with or without disabilities

Exclusion Criteria:

* Second Life: People with disabilities - does not include those without disabilities or clinicians from Second Life.
* Second Life: People without disabilities - does not include those with disabilities or clinicians from Second Life.
* Second Life: clinicians - does not include those with or without disabilities from Second Life.
* Urban: does not include clinicians

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Both: both female and male participants are being studied
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hillary R Bogner, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Vries McClintock HF, Barg FK, Katz SP, Stineman MG, Krueger A, Colletti PM, Boellstorff T, Bogner HR. Health care experiences and perceptions among people with and without disabilities. Disabil Health J. 2016 Jan;9(1):74-82. doi: 10.1016/j.dhjo.2015.08.007. Epub 2015 Sep 5. PMID 26482010
- [Result] Bogner HR, de Vries McClintock HF, Hennessy S, Kurichi JE, Streim JE, Xie D, Pezzin LE, Kwong PL, Stineman MG. Patient Satisfaction and Perceived Quality of Care Among Older Adults According to Activity Limitation Stages. Arch Phys Med Rehabil. 2015 Oct;96(10):1810-9. doi: 10.1016/j.apmr.2015.06.005. Epub 2015 Jun 26. PMID 26119464

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Second Life: People With Disabilities | Second Life: People Without Disabilities | Second Life: Clinicians | Urban Group
Started | 23 | 10 | 6 | 10
Completed | 23 | 10 | 6 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Second Life: People With Disabilities | Second Life: People Without Disabilities | Second Life: Clinicians | Urban Group | Total
Number analyzed (Participants) | 23 | 10 | 6 | 10 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 5 | 4 | 3 | 27
  >=65 years | 8 | 5 | 2 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43 (8.2) | 45 (6.3) | 56 (2.7) | 68 (7.9) | 59 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 8 | 4 | 8 | 40
  Male | 3 | 2 | 2 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 2 | 6
  Not Hispanic or Latino | 21 | 8 | 6 | 8 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 0 | 4 | 11
  White | 14 | 2 | 6 | 4 | 26
  More than one race | 5 | 3 | 0 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 10 | 6 | 10 | 49
Number of people analyzed in each focus group [Count of Participants; unit: Participants] | 23 | 10 | 6 | 10 | 49

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Medical Care Survey
Description: Multinomial logistic regression models will be used to determine the degree to which people with disabilities and without have satisfaction with medical care obtained from the survey. The scale ranges from 1 (not satisfied) to 4 (very satisfied) with their medical care. Higher scores represent more satisfaction with medical care. Unit of measurement is units on a scale.
Time Frame: One year
Population: Satisfaction with healthcare
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Second Life: People Without Disabilities: People without disabilities recruited fro the virtual world Second Life
- Second Life: Clinicians: Clinicians recruited from the virtual world Second life
- Urban: People with and without disabilities recruited from an Urban community
Arm/Group | Second Life: People With Disabilities | Second Life: People Without Disabilities | Second Life: Clinicians | Urban
Number analyzed (Participants) | 23 | 10 | 6 | 10
units on a scale | 3.4 (1.2) | 3.8 (1.7) | 3.6 (1.9) | 3.0 (2.9)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Second Life:People Without Disabilities: People without disabilities recruited from the virtual world, Second life.
Arm/Group | Second Life: People With Disabilities | Second Life:People Without Disabilities | Second Life: Clinicians | Urban
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/10 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/10 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 0/23 | 0/10 | 0/6 | 0/10

LIMITATIONS AND CAVEATS:
The qualitative nature of this study does not provide insight for causal inferences. Second, the small number of participants limits this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (6):
  • Informed Consent Form: clinician (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT02626910/ICF_000.pdf
  • Informed Consent Form: PWD_SL (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT02626910/ICF_001.pdf
  • Informed Consent Form: PWD_URBAN (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT02626910/ICF_002.pdf
  • Informed Consent Form: PWOD_SL (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT02626910/ICF_003.pdf
  • Informed Consent Form: PWOD_URBAN (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT02626910/ICF_004.pdf
  • Study Protocol and Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT02626910/Prot_SAP_005.pdf